CLINICAL TRIAL: NCT01509118
Title: Rivaroxaban Safety Profile in the Prophylaxis of Venous Thromboembolism After Hip Fracture Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Collaborators: Chulalongkorn University (Other); Chiang Mai University (Other); Thammasat University (Other); Police General Hospital (Other); Saint Louis Hospital,bangkok,Thailand (Unknown); Bhumibol Adulyadej Hospital (Other)
Responsible Party: Principal Investigator, Dr.Thanainit Chotanaphuti, Colonel, Phramongkutklao College of Medicine and Hospital
Other Study IDs: 15635
Record Dates: First submitted 2012-01-08; First posted 2012-01-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Open Fracture of Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Arterial and venous thromboembolism represents one of the most common preventable health problems. Patients undergoing surgery, especially hip fracture surgery are at high risk for deep vein thromboembolism (VTE) without thromboprophylaxis. In the absence of prophylaxis, the incidence of fatal pulmonary embolism (PE) after Hip Fracture Surgery (HFS) is reportedly 4%-12%. Provision of thromboprophylaxis to all patients who undergo HFS is recommended.

DETAILED DESCRIPTION:
Rivaroxaban is the first agent of a new class of drugs acting as direct factor Xa inhibitors with oral bioavailability. Highly selective inhibition of factor Xa by rivaroxaban is expected to inhibit the amplified burst of thrombin generation and may result in more effective inhibition of thrombus formation with a favorable safety profile. In Thailand rivaroxaban is indicated for the prevention of VTE in patients undergoing major orthopedic surgery of the lower limbs including surgery for hip fractures. There are limited number of observational studies of rivaroxaban in thromboembolism after hip fracture surgery as the approved indication in most countries are for thromboprophylaxis in hip and knee arthroplasty. The broader indications and the high number of hip fracture surgeries in Thailand allow us to explore a pattern of safety profile particularly bleeding complications and risk factors in patients receiving rivaroxaban thromboprophylaxis after hip fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years old in men or post-menopause in women
* Patients, who are undergoing standard surgery for fracture of the upper third of the femur, including femoral head, neck, trochanteric and sub-trochanteric fracture and the surgery is planned within 7 days after admission
* Patients, who are eligible for thromboprophylaxis. Such patients will be enrolled only after physician's decision to prescribe rivaroxaban for thromboprophylaxis has been made. The decision is totally based on standard of medical practice.
* Patients, who agree to participate, return to follow-up visits, and who have signed informed consent to participate in the study.

Exclusion Criteria:

* Trauma affecting more than 1 organ system
* Pathological fracture secondary to malignant disease
* Clinically significant bleeding excluding drainage
* Documented congenital or acquired bleeding disorder
* Patients, who have contraindications for thromboprophylaxis or contraindications to take rivaroxaban according to FDA-approved product label
* Patient on oral anticoagulation therapy in the past 7 days
* Pregnancy or breastfeeding
* Patients who are simultaneously participating in a different study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rivaroxaban safety profile will be observed in 500 patients
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Thanainit Chotanaphut, M.D., Principal Investigator — Department of Orthopaedic Surgery Pharmongkutklao Hospital
Locations (7):
- Thailand (7):
  - Orthopedic/Board of Orthopedic Surgery, Saint Louis Hospital, Bangkok, Bangkok
  - Department of Orthopedic Surgery, Bhumibol Adulyadej Hospital, Bangkok, Bangkok
  - Department of Orthopaedics, Chulalongkorn Hospital, Pathumwan, Bangkok
  - Department of Orthopedic Surgery, Police General Hospital, Pathumwan, Bangkok
  - Department of Orthopaedic surgery Pharmongkutklao Hospital, Rajathevee, Bangkok
  - Department of Orthopaedics, Thammasat University, Klong Luang, Changwat Pathum Thani
  - Department of Orthopaedic Surgery,Chiang Mai University, Muang, Chiang Mai